CLINICAL TRIAL: NCT00293761
Title: A Study of Glaucoma Therapy to Treat Open-Angle Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C-05-51
Record Dates: First submitted 2006-02-17; First posted 2006-02-20 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2012-03

CONDITIONS: Open-angle Glaucoma; Ocular Hypertension
Keywords: open-angle; glaucoma; ocular; hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension; Glaucoma; Hypertension | interventions — Travoprost

ARMS (2):
- Travatan, Investigational (Experimental)
  Interventions: Drug: Travoprost, Investigational
- Travatan (Active Comparator)
  Interventions: Drug: Travoprost (TRAVATAN)

INTERVENTIONS:
Drug: Travoprost, Investigational — One drop in study eye once daily for 13 days
  Arms: Travatan, Investigational
Drug: Travoprost (TRAVATAN) — One drop in study eye once daily for 13 days
  Other Names: TRAVATAN
  Arms: Travatan

SUMMARY:
The purpose of the study is to determine whether a glaucoma therapy is safe and effective in treating patients with open-angle glaucoma or ocular hypertension

ELIGIBILITY:
Inclusion Criteria:

* Adult patients of either sex of any race diagnosed with open-angle glaucoma (with or without pseudoexfoliation or pigment dispersion component) or ocular hypertension.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Under age 18.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2006-01; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Mean IOP

REFERENCES:
- [Result] Gross RL, Peace JH, Smith SE, Walters TR, Dubiner HB, Weiss MJ, Ochsner KI. Duration of IOP reduction with travoprost BAK-free solution. J Glaucoma. 2008 Apr-May;17(3):217-22. doi: 10.1097/IJG.0b013e31815a3472. PMID 18414108